CLINICAL TRIAL: NCT05836597
Title: Effectiveness and Safety of Virtual Reality for the Treatment of Functional Dyspepsia
Brief Title: Functional Dyspepsia Treatment Using Virtual Reality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David J. Cangemi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-001973
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental (Experimental): Experimental VR
  Interventions: Device: Virtual reality
- Sham (Sham Comparator): Sham VR
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — Virtual reality

SUMMARY:
The purpose of this study is to evaluate the effectiveness of using virtual reality to treat gastrointestinal symptoms related to functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of dyspepsia thought to represent functional dyspepsia, meeting Rome IV criteria
* Had an upper endoscopy and assessment for Helicobacter pylori; if a patient is found to have H. pylori, treatment with confirmed eradication (by stool antigen test or urea breath test) will be required before the patient is eligible for study inclusion.
* Patients will be considered for the study if they have undergone a complete history and physical examination during a previously scheduled consultation/evaluation visit with a gastroenterologist in the Mayo Clinic Florida General GI or Motility clinic.

Exclusion Criteria:

* Symptoms are thought to represent an organic disorder (e.g., peptic ulcer disease, hepatitis, pancreatitis, inflammatory bowel disease, type I diabetes, a known malignancy, radiation-induced injury, an active infection, vasculitis, celiac disease), or patients have known uncontrolled GERD, esophagitis, eosinophilic esophagitis, or untreated H. pylori.
* Patients with gastroparesis or cyclic vomiting syndrome.
* Patients with prior surgery to the esophagus, stomach or duodenum.
* Patients taking opioids.
* Patients with motion sickness, vertigo, or a seizure disorder
* IBS symptoms are not predominant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in abdominal pain scores | Baseline, 8 weeks
  Measured by the Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) questionnaire individual scores for abdominal pain. Scored 0-5, with higher scores representing more severe symptoms.

SECONDARY OUTCOMES:
Overall PAGI-SYM scores | Baseline, 8 weeks
  Measured by the Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) questionnaire. All symptoms scored 0-5, with higher scores representing more severe symptoms. A total PAGI-SYM score is determined by calculating the average of all symptom scores
Change in nausea/vomiting | Baseline, 8 weeks
  Measured by the Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) questionnaire individual scores for nausea/vomiting. Scored 0-5, with higher scores representing more severe symptoms.
Change in bloating | Baseline, 8 weeks
  Measured by the Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) questionnaire individual scores for bloating. Scored 0-5, with higher scores representing more severe symptoms.
Change in post-prandial fullness | Baseline, 8 weeks
  Measured by the Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) questionnaire individual scores for early satiety/postprandial fullness. Scored 0-5, with higher scores representing more severe symptoms.
Change in heartburn | Baseline, 8 weeks
  Measured by the Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) questionnaire individual scores for heartburn. Scored 0-5, with higher scores representing more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: David Cangemi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials